CLINICAL TRIAL: NCT05128799
Title: Effect of the 3 Wishes Program on Bereaved Families' End-of-Life Care Perceptions
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Thanh H. Neville, MD, MSHS, Associate Professor, University of California, Los Angeles
Other Study IDs: Effect of 3WP on BFS
Record Dates: First submitted 2021-11-10; First posted 2021-11-22 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: End of Life; Death
Keywords: end of life; palliative care; intensive care unit
MeSH Terms: conditions — Death

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 3WP: Patients who had 3WP as part of their end-of-life care
  Interventions: Other: 3 Wishes Program (3WP)
- Usual Care: Patients who did not have 3WP as part of their end-of-life care

INTERVENTIONS:
Other: 3 Wishes Program (3WP) — The 3 Wishes Program (3WP) is a palliative care intervention in which small wishes are implemented by healthcare workers (HCWs) in an effort to improve the EOL experience for dying patients and their families. Examples of wishes include playing the patient's favorite music, providing a non-hospital blanket, orchestrating a final "date night," decorating a patient's room to reflect their identify, and providing grieving family members with keepsakes such as thumbprint keychains, framed EKG mementos, or word clouds.
  Groups: 3WP

SUMMARY:
Dying in the intensive care unit (ICU) can be a source of trauma for patients and their families. The 3 Wishes Program is a palliative care initiative in which healthcare workers fulfills small wishes to provide a personalized, humanizing experience at the end of life (EOL) for dying patient and their families. The investigators' objective is to assess families' ratings of EOL care for ICU decedents who received the 3WP as part of their EOL care versus usual care.

DETAILED DESCRIPTION:
This is a quality improvement study to evaluate the effect of the 3 Wishes Program (3WP) on end-of-life (EOL) care in the adult ICUs of a two-hospital academic healthcare system.

At this health system, patients were invited to participate in the 3WP once a decision to withdraw life support was made or the health care team agreed that the patient's probability of dying in the hospital or on discharge to hospice was >95%. As a quality improvement measure, 3WP initiation was up to the discretion of the clinical team. Patients and/or families provide verbal consent. HCWs, mostly nurses, asked how they might bring comfort to a dying patient and their family in the final hours or days of life. Wishes can also be suggested by the clinical team.

A modified Bereaved Family Survey (BFS), a cover letter and a self-addressed stamped envelope were mailed to the next of kin three months after the patient's death. Surveys had no identifying information and were tracked using a unique code. No incentive was offered. Two weeks following the initial mailing, non-responders received up to three telephone calls (at least one attempt after 5PM and maximum two voice messages) to request the return of the survey or to complete it by telephone, if preferred.

BFS results were compared between patients who received the 3WP and those who did not. Demographics and clinical characteristics were abstracted and included in multivariate models.

ELIGIBILITY:
Inclusion Criteria:

* For participation in the 3WP, if there was a decision to withdraw life support or the health care team agreed that the patient's probability of dying in the hospital or on discharge to hospice was >95%
* For surveys, next of kin/surrogate of a patient who died in the ICU during the study period
* For surveys, speaks English

Exclusion Criteria:

* <21 years old
* does not speak English

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who died in the adult ICU and their families
Sampling Method: Non-Probability Sample
Enrollment: 314 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2021-07-04 (Actual); Study Completion 2021-11-09 (Actual)

PRIMARY OUTCOMES:
Emotional and Spiritual Support | 3 months after the patient's death
  Emotional and spiritual support factor score on the Bereaved Family Survey total score ranges 0-9 (higher is better)

SECONDARY OUTCOMES:
Bereaved Family Survey Performance Measure | 3 months after the patient's death
  overall assessment of quality of end of life care 0-1 (higher is better)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UCLA Santa Monica Medical Center, Santa Monica, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vanstone M, Neville TH, Clarke FJ, Swinton M, Sadik M, Takaoka A, Smith O, Baker AJ, LeBlanc A, Foster D, Dhingra V, Phung P, Xu XS, Kao Y, Heels-Ansdell D, Tam B, Toledo F, Boyle A, Cook DJ. Compassionate End-of-Life Care: Mixed-Methods Multisite Evaluation of the 3 Wishes Project. Ann Intern Med. 2020 Jan 7;172(1):1-11. doi: 10.7326/M19-2438. Epub 2019 Nov 12. PMID 31711111
- [Background] Neville TH, Bear DK, Kao Y, Xu XS, Hjelmhaug K, Quebral D, Sanaee N, Hainje J, Arriola G, Granone MC, White E, Chaturvedi A, Yu S, Clarke F, Cook DJ. End-of-Life Care During the Coronavirus Disease 2019 Pandemic: The 3 Wishes Program. Crit Care Explor. 2021 Oct 8;3(10):e549. doi: 10.1097/CCE.0000000000000549. eCollection 2021 Oct. PMID 34651136
- [Background] Vanstone M, Sadik M, Smith O, Neville TH, LeBlanc A, Boyle A, Clarke FJ, Swinton ME, Takaoka A, Toledo F, Baker AJ, Phung P, Cook DJ. Building organizational compassion among teams delivering end-of-life care in the intensive care unit: The 3 Wishes Project. Palliat Med. 2020 Oct;34(9):1263-1273. doi: 10.1177/0269216320929538. Epub 2020 Jun 10. PMID 32519615
- [Background] Neville TH, Clarke F, Takaoka A, Sadik M, Vanstone M, Phung P, Hjelmhaug K, Hainje J, Smith OM, LeBlanc A, Hoad N, Tam B, Reeve B, Cook DJ. Keepsakes at the End of Life. J Pain Symptom Manage. 2020 Nov;60(5):941-947. doi: 10.1016/j.jpainsymman.2020.06.011. Epub 2020 Jun 21. PMID 32574658